CLINICAL TRIAL: NCT06111209
Title: A Pilot Study to Evaluate the Anabolic Effect of Testosterone on Muscles of the Pelvic Floor in Older Women With Stress Urinary Incontinence
Brief Title: The Anabolic Effect of Testosterone on Pelvic Floor Muscles
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P002632; R01DK136904 (NIH)
Record Dates: First submitted 2023-10-18; First posted 2023-11-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence; Menopause
Keywords: stress urinary incontinence; testosterone therapy; menopause; pelvic floor disorders
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Floor Disorders | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Active Comparator): Testosterone Cypionate 25-mg weekly by intramuscular injection
  Interventions: Drug: Testosterone cypionate
- Placebo (Placebo Comparator): Placebo intramuscular injections weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone cypionate — weekly by intramuscular injection
  Arms: Testosterone
Drug: Placebo — weekly by intramuscular injection
  Arms: Placebo

SUMMARY:
Stress urinary incontinence is the most common female pelvic floor disorder encountered in clinical practice with significant negative impact on quality of life. The prevalence of urinary incontinence increases with aging, and weakness of the pelvic floor muscles contributes to the development of stress urinary incontinence. Given that androgen receptors are expressed throughout the pelvic floor, the anabolic effects of androgens on pelvic floor muscles may provide a therapeutic option in women with stress urinary incontinence. The investigators are conducting a randomized, double-blind, placebo-controlled proof-of-concept trial in older postmenopausal women with stress urinary incontinence to assess whether testosterone therapy can increase pelvic floor muscles and improve urinary function.

DETAILED DESCRIPTION:
The investigators are conducting a 12-week double-blind, randomized-controlled, proof-of-concept pilot trial to determine the anabolic effect of testosterone therapy on pelvic floor muscles in postmenopausal women, 60 years and older, with stress urinary incontinence. The first aim is to compare the efficacy of testosterone supplementation versus placebo on the volume of levator ani muscles of the pelvic floor, assessed by magnetic resonance imaging (MRI). The second aim is to assess the efficacy of testosterone supplementation in improving indices of urodynamic function (i.e., bladder, urethra, and sphincter function), assessed by urodynamic testing. These urodynamic measures include Valsava leak point pressure, urethral pressure profile, cystometry and electromyography. As an exploratory aim, the efficacy of testosterone treatment relative to placebo will be assessed using self-reported urinary symptoms assessed by the Urogenital Distress Inventory (UDI) and quality of life assessed by the Incontinence Impact Questionnaire (IIQ).

ELIGIBILITY:
Inclusion Criteria:

* Women, age 60 years and older.
* Medically documented pure stress urinary incontinence on physical exam or urodynamic testing.
* Normal mammogram within the last 12 months
* Endometrial thickness of ≤4 mm in women with an intact uterus assessed by endometrial ultrasound.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* • Medically documented urge or mixed urinary incontinence (stress and urge) on physical exam or urodynamic testing.

  * Participating in pelvic floor muscle training (PFMT) therapy currently or in the past 3 months
  * Previous pelvic surgery (i.e., hysterectomy, pelvic organ prolapse repair, mid-urethral sling placement, injection of urethral bulking agents) or radiation treatment to the pelvis.
  * History of ≥ Grade 3 pelvic organ prolapse
  * Neurologic disorder causing UI or bladder dysfunction (i.e., multiple sclerosis, Parkinson's disease, stroke, cerebral palsy, spinal cord injury)
  * Current urinary tract infection
  * History of breast or endometrial cancer
  * Use of systemic estrogen therapy in the past 3 months
  * Baseline hematocrit >48%, serum creatinine >2.5 mg/dL; HbA1c >8.0%; BMI >40 kg/m2
  * Uncontrolled hypertension defined as an average of two blood pressure readings of greater than 160/100.
  * Subjects who are on insulin therapy will be excluded.
  * Uncontrolled congestive heart failure
  * Myocardial infarction, acute coronary syndrome, revascularization surgery or stroke within 6 months
  * History of pulmonary embolism, deep vein thrombosis or a genetic thromboembolic disorder
  * History of bipolar disorder, schizophrenia or untreated major depression
  * Presence of metallic implants (pacemakers, aneurysm clips, etc.) that preclude the patient from undergoing MRI

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in pelvic floor muscle volume | 12 weeks
  volume of levator ani muscles of the pelvic floor, assessed by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Change in abdominal leak point pressure | 12 weeks
  abdominal leak point pressure will be measured by a urodynamic function study
Change in urine flow rate | 12 weeks
  urine flow rate will be measured by urodynamic function a study
Change in bladder pressure | 12 weeks
  bladder pressure will be measured during filling, storage and voiding by urodynamic study
Change in post void residual urine volume | 12 weeks
  post void residual urine volume will be measured using bladder ultrasound
Change in urinary symptoms | 12 weeks
  self-reported urinary symptoms will be assessed by the Urogenital Distress Inventory (UDI). Total score ranges from 6-24 with higher scores indicating higher severity of symptoms
Change in quality of life | 12 weeks
  quality of life will be assessed by the Incontinence Impact Questionnaire (IIQ). Total score ranges from 0-21 with higher scores indicating worse impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Huang, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No